CLINICAL TRIAL: NCT07203625
Title: Intravenous Tenecteplase Before Interhospital Transfer for Thrombectomy in Acute Basilar Artery Occlusion at 4.5 to 24 Hours
Brief Title: Tenecteplase Before Interhospital Transfer in Acute Basilar Artery Occlusion at 4.5 to 24 Hours
Acronym: OPTION-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XMEC-2025-003
Record Dates: First submitted 2025-09-16; First posted 2025-10-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke; Basilar Artery Occlusion
Keywords: basilar artery occlusion; thrombolysis; interhospital transfer
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Patients will receive intravenous Tenecteplase 0.25 mg/kg body-weight up to a maximum of 25mg before the transfer. A single bolus dose should be administered over 5-10 seconds based on patient weight. Transfer to ECCs for thrombectomy should be initiated immediately after Tenecteplase administration.
  Interventions: Drug: Tenecteplase thrombolysis
- Control group (No Intervention): Patients will be directly transferred to ECCs for thrombectomy according to Chinese Guidelines for Diagnosis and Treatment of Acute Ischemic Stroke 2023.

INTERVENTIONS:
Drug: Tenecteplase thrombolysis — Patients will receive intravenous Tenecteplase 0.25 mg/kg body-weight up to a maximum of 25mg before the transfer. A single bolus dose should be administered over 5-10 seconds based on patient weight. Transfer to ECCs for thrombectomy should be initiated immediately after Tenecteplase administration.
  Other Names: rhTNK-tPA
  Arms: Interventional group

SUMMARY:
This study is designed to investigate the efficacy and safety of intravenous tenecteplase before interhospital transfer from a non-endovascular capable center(nECC) to an endovascular capable center (ECC) for thrombectomy in patients with acute ischemic stroke (AIS) caused by neuroimaging-confirmed acute basilar artery occlusion (BAO) between 4.5-24 hours of symptom onset.

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-label, blinded endpoint (PROBE), randomized controlled trial in patients with acute ischemic stroke due to BAO first presenting to a nECC and intending to undertake thrombectomy in an ECC.

Patients will be required to have occlusion of the basilar artery on baseline computed tomography angiography (CTA)/magnetic resonance angiography (MRA) at the nECC. Patients will be randomized to either intravenous tenecteplase (0.25mg/kg, maximum 25mg)or not before interhospital transfer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years; 2. Patients presenting with posterior circulation ischemic stroke symptoms due to BAO; 3. BAO confirmed by computed tomographic angiography (CTA)/ magnetic resonance angiography (MRA); 4. Time from symptom onset to randomization within 4.5-24 hours, stroke onset is defined as the time the patient was last known to be well (including wake-up stroke and unwitnessed stroke); 5. Baseline National Institute of Health Stroke Scale (NIHSS) score obtained prior to randomization ≥6; 6. Functionally independent (modified Rankin Scale [mRS] 0-2) prior to stroke onset; 7 Intended to transfer to CSCs for thrombectomy 8. Written informed consent from patients or legally responsible representatives

Exclusion Criteria:

* 1 Posterior Circulation Acute Stroke Prognosis Early CT score (PC-ASPECTS) < 6 on computed tomography (CT)/CTA-Source Images/MRI with diffusion-weighted imaging (DWI) 2 CT/MR shows evidence of intracranial hemorrhage and tumor (except small meningioma) 3 Complete cerebellar infarct on CT/MRI with significant mass effect and compression of the 4th ventricle 4 Bilateral extensive brainstem infarction on CT/MRI 5 Simultaneous occlusion of both anterior and posterior circulation confirmed by CTA/MRA/DSA (patients with a history of occlusion of anterior circulation can be included) 6 Treatment with a thrombolytic within the last 72 hours or intention to receive intravenous thrombolysis 7 Known hypersensitivity or allergy to any ingredients of Tenecteplase 8 Any other contra-indication for intravenous thrombolysis except for the time criteria 9 Known hereditary or acquired hemorrhagic diathesis 10 Impairment in coagulation due to comorbid disease or anticoagulant use. If on warfarin, international normalized ratio (INR) >1.7 or prothrombin time >15s; if use of any direct oral anticoagulant within the last 48 hours; if use of heparin/heparinoid within the last 24 hours 11 Ischemic stroke or myocardial infarction in previous 3 months 12 Previous intracranial hemorrhage, active internal bleeding (gastrointestinal or urinary tract hemorrhage) in previous 3 months 13 Severe, uncontrolled hypertension (systolic blood pressure >185mmHg or diastolic blood pressure >110mmHg) 14 Baseline blood glucose <50mg/dl or >400mg/dl 15 Baseline platelet count <100,000/μL 16 Undergoing hemodialysis or peritoneal dialysis; known severe renal insufficiency with glomerular filtration rate <30mL/min or serum creatinine >220mmol/L (2.5mg/dL) 17 Known severe, life-threatening allergy (more severe than skin rash) to contrast agents 18 Patients with acute stroke within the first 48 hours after percutaneous cardiac, cerebrovascular interventions and major surgery 19 Known diagnosis or clinical suspicion of cerebral vasculitis 20 Known diagnosis or clinical suspicion of endocarditis 21 Pregnancy or lactating; 22 Other serious, advanced or terminal illness with life expectancy less than 6 months 23 Current participation in any investigational study that may confound outcome assessment of the study 24 Any condition that, in the judgement of the investigator, is inappropriate for participation in the trial or could impose hazards to the patient (e.g. inability to understand and/or follow the study procedures and/or follow-up due to mental disorders, cognitive or emotional disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dichotomized mRS of 0-2 vs. 3-6 | 90±7 days
  Dichotomized mRS of 0-2 vs. 3-6 at 90±7 days; modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

SECONDARY OUTCOMES:
Ordinal mRS score | 90 (±7) days
  Ordinal mRS score at 90 (±7) days; modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Dichotomized mRS of 0-1 vs. 2-6 | 90 (±7) days
  Dichotomized mRS of 0-1 vs. 2-6 at 90 (±7) days
Dichotomized mRS of 0-3 vs. 4-6 | 90 (±7) days
  Dichotomized mRS of 0-3 vs. 4-6 at 90 (±7) days
Early dramatic clinical response rate | 24 (±12) hours
  Early dramatic clinical response rate at 24 (±12) h, defined as a NIHSS score of 0 or 2 or NIHSS drop of ≥8 from baseline
Arterial recanalization during interhospital transfer | At ECC before thrombectomy
  Arterial recanalization during interfacility transfer, evaluated with the angiography (CTA/MRA/first run of DSA) at ECC, and rated on the arterial occlusive lesion (AOL)
Successful reperfusion | At end-of-procedure angiography
  Successful reperfusion at end-of-procedure angiography, defined as expanded Treatment in Cerebral Infarction (eTICI) score of 2b, 2c, or 3 on angiography
First pass reperfusion | Immediately after the thrombectomy
  First pass reperfusion defined as eTICI 2c or greater after the first thrombectomy pass
Arterial recanalization | 24(±12) hours
  Arterial recanalization at 24(±12)h, evaluated with CTA/MRA and rated on the AOL
EQ-5D-5L | 90 (±7) days
  Score on the EQ-5D-5L at 90 (±7) days;(EQ-5D-5L: Minimum Score 5, Maximum score 25, lower scores mean a better quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No